CLINICAL TRIAL: NCT02890173
Title: A Double Blind Study of CS-3150 to Evaluate Efficacy and Safety Compared to Eplerenone in Patients With Essential Hypertension (ESAX-HTN Study)
Brief Title: Study of CS-3150 in Patients With Essential Hypertension
Acronym: ESAX-HTN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS3150-A-J301
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2017-08

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Mineralocorticoid receptor antagonist; Esaxerenone; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Essential Hypertension | interventions — esaxerenone; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CS-3150 2.5 mg (Experimental): CS-3150 2.5 mg, orally, once daily after breakfast for 12 weeks
  Interventions: Drug: CS-3150
- CS-3150 5.0 mg (Experimental): CS-3150 5 mg, orally, once daily after breakfast for 12 weeks
  Interventions: Drug: CS-3150
- Eplerenone (Active Comparator): Eplerenone 50 mg, orally, once daily after breakfast for 12 weeks
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: CS-3150
  Arms: CS-3150 2.5 mg; CS-3150 5.0 mg
Drug: Eplerenone
  Other Names: Inspra
  Arms: Eplerenone

SUMMARY:
To evaluate antihypertensive effect and safety of CS-3150 compared to Eplerenone in patients with essential hypertension.

DETAILED DESCRIPTION:
Primary objective is to evaluate antihypertensive effect and safety of CS-3150 2.5 mg compared to Eplerenone in patients with essential hypertension.

Secondary objective is to evaluate antihypertensive effect and safety of CS-3150 5.0 mg compared to 2.5 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 years or older at informed consent
* Subjects with essential hypertension satisfying the following blood pressure criteria;

  * Sitting SBP: ≥ 140 mmHg and < 180 mmHg
  * Sitting DBP: ≥ 90 mmHg and < 110 mmHg
  * Mean 24 hr BP: SBP ≥ 130 and DBP ≥ 80 mmHg

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Diabetic nephropathy or diabetes mellitus with albuminuria
* Serum potassium level < 3.5 or ≥ 5.1 mEq/L
* Reversed day-night life cycle including overnight workers
* eGFR < 60 mL/min/1.73 m^2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting blood pressure | Baseline to end of Week 12
  Change from baseline in sitting systolic (SBP) and diastolic blood pressure (DBP).

SECONDARY OUTCOMES:
Change from baseline in 24 hour average blood pressure | Baseline to end of Week 12
  Change from baseline in 24 hour average systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo Co., Ltd.
Locations (1):
- Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Ito S, Itoh H, Rakugi H, Okuda Y, Yoshimura M, Yamakawa S. Double-Blind Randomized Phase 3 Study Comparing Esaxerenone (CS-3150) and Eplerenone in Patients With Essential Hypertension (ESAX-HTN Study). Hypertension. 2020 Jan;75(1):51-58. doi: 10.1161/HYPERTENSIONAHA.119.13569. Epub 2019 Dec 2. PMID 31786983